CLINICAL TRIAL: NCT06819449
Title: Rab 32 Gene Polymorphisms as a Prognostic Factor in Leprosy Patients and Its Relation to Multiple Drug Therapy: Randomized Clinical Trial
Brief Title: Rab 32 Gene Polymorphisms as a Prognostic Factor in Leprosy Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Lydia Atef Nassief, Resident of Dermatology , venereology and andrology at Faculty of medicine, South Valley University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Rab 32 gene polymorphisms
Record Dates: First submitted 2025-01-21; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-12

CONDITIONS: Leprosy; Mycobacterium Leprae Infection
MeSH Terms: conditions — Leprosy | interventions — Dapsone; Clofazimine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Leprosy Patients (Active Comparator): About 40 patients suffering from Leprosy and will treated by Multi drug therapy as ( dapsone _ clofazimine _ rifampcin) then to assess the role of Rab 32 gene.by taking Two millimetres of venous blood from each participant At the end of third month therapy.
  Interventions: Drug: Dapsone
- Group B: Healthy People (Active Comparator): About 10 Healthy People. no drugs used and then to assess the role of Rab 32 gene.by taking Two millimetres of venous blood from each participant
  Interventions: Drug: Dapsone

INTERVENTIONS:
Drug: Dapsone — To evaluate the effect of the multi drug therapy in leprotic patients and their side effects and to assess the role of Rab 32 gene in leprosy prognosis and to know its association with the multi drug therapy.
  Other Names: clofazimine; rifampcin

SUMMARY:
Mycobacterium leprae is a slow-growing bacillus that causes leprosy. the infection may take two to ten years to incubate. While the exact mechanism of infection transmission is unknown, direct bacillus absorption through the nasal or respiratory mucosa and aerosolized nasal secretions are the most common theories. The bacteria is subsequently transported by the bloodstream to the peripheral nerves, where it can result in tissue damage from painless burns and ulcers as well as irreparable nerve damage that results in a loss of protective feeling.

DETAILED DESCRIPTION:
One of the most common host cells that mycobacteria encounter is macrophages. The process of monocyte-derived macrophages phagocytosing M. leprae is controlled by protein kinase and can be facilitated by complement receptors CR1 (CD35), CR3 (CD11b/CD18), and CR4 (CD11c/CD18). A Th2 cytokine profile appears to be correlated with nonreactivity to M.Leprea.

The Ridley-Jopling classification (1962) divides leprosy into six forms: Tuberculoid (TT), Borderline Tuberculoid (BT), Borderline-borderline Mid-borderline (BB), Borderline-Lepromatous (BL), Subpolar Lepromatous (LLs), and Polar Lepromatous (LLp). These categories are based on clinical, histopathological, and immunological criteria. According to WHO, leprosy is classified into two groups: the paucibacillary (PB) and multibacillary (MB) types, to aid in treatment.

Leprosy is treated as an outpatient procedure using WHO-standardized regimens from 1982, which essentially consist of three first-line medications: clofazimine, rifampicin, and dapsone. This relationship is referred to as polychemotherapy, or MDT (PCT). With minimal bactericidal activity, sulfone (diaminodiphenyl sulfone, or DDS), commonly referred to as dapsone, primarily acts as a bacteriostatic agent.

It most likely functions as an antagonist of para- aminobenzoic acid (PABA), preventing M. leprae from using it to synthesize folic acid. It is well-tolerated and has a number of adverse effects, most of which do not require stopping treatment.

The primary bactericidal effect of rifampicin (RMP), a semi-synthetic derivative of rifamycin B, is observed. It functions by preventing the RNA-polymerase enzyme in the bacillus from growing. RMP has been used to treat leprosy since 1963. Most of the bacilli become non-viable after a few days of therapy, and its use is crucial in all clinical types of leprosy. Clofazimine (CLF) is an iminophenazine dye . It has a mild bactericidal action, acting slowly on M. leprae and destroying 99% of the bacteria in approximately five months. Its efficacy is similar to DDS. CLF has an important anti-inflammatory action.

With an estimated heritability of up to 57%, family studies and community epidemiological surveys have amply established the significant role that host genetics plays in an individual's vulnerability to leprosy.

RAB32 is a low molecular weight G protein belonging to the Ras superfamily. It is necessary for the production of autophagic vacuoles and the control of autophagy's removal of aggregated proteins. Rab32 may play a similar role in the pathogenesis of leprosy, according to a recent study that found the protein controls the recruitment of cathepsin D to phagosomes containing Mycobacterium tuberculosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes with positive slit skin smear for m.leprae .

Exclusion Criteria:

* Contraindications to Multi drug therapy :
* Patients with hypersensitivity to sulfa .
* Patients with hypersensitivity to clofazimine or rifampcin.
* pregnant or lactating women.

Ages: 5 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2025-12-10 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Treatment of leprosy | 6 Months
  About 40 of Participants With Treatment-Related Adverse Events as Assessed by measuring the of Rab 32 gene ( Rs2275606 ) polymorphism using real time PCR for Evaluation of the multi drug therapy on Leprotic Patients

CONTACTS AND LOCATIONS:
Overall Officials: Eisa Mohammed Hegazy, Assist. Prof, Study Chair — Dermatology, Venereology and Andrology. Faculty of Medicine,South Valley University
Locations (1):
- Qina University hospital, South Valley University Hospital, Qina, Egypt